CLINICAL TRIAL: NCT04947098
Title: Prevent Cancer-Greenville: A Center for Cancer Prevention and Wellness Research Project
Brief Title: Prevent Cancer- Greenville
Acronym: CCPW
Status: Recruiting | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00077309
Record Dates: First submitted 2021-04-29; First posted 2021-07-01 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cancer; High-Risk Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and cheek swab specimens will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prevent Cancer-Greenville was created to provide individuals with the opportunity to have their risk of developing cancer studied. Some individuals may be at a higher risk due to their personal lifestyle, family history and/or exposures. If subjects are found to be at high risk for developing a disease, they will be sent to a healthcare provider for further care.

DETAILED DESCRIPTION:
Participants' personal history, lifestyle behaviors and blood, urine, and cheek swab specimens will be used to detect changes or trends that might put them at risk for developing cancer. Some individuals may be at an above average risk of cancer due to lifestyle, family background, personal genetic makeup, or environmental exposures. This will be determined by a process called risk stratification. Risk stratification involves looking at all health-related aspects of a person, determining their individualized risk through screening, and educating them on measures to reduce potential for disease. Participants will complete a yearly health assessment which includes measurements for nutrition, activity, individual risk factors and body composition, including weight height and a special scale which measures fluid and fat.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2028-11-08 (Estimated); Study Completion 2029-11-08 (Estimated)

PRIMARY OUTCOMES:
Assess changes in nutrition by nutrition questionnaire | Yearly follow up for 10 years
  Nutrition will be assessed yearly by a questionnaire based on nutrition recommendations from the American Institute for Cancer Research and the U.S. Department of Health and Human Services.
Assess changes in physical activity by physical activity questionnaire | Yearly follow up for 10 years
  Physical activity will be assessed yearly a questionnaire based on physical activity recommendations from the U.S. Department of Health and Human Services.
Assess changes in smoking habits | Yearly follow up for 10 years
  Participants will be educated on healthy lifestyle habits and smoking habits will be assessed yearly.
Assess changes in alcohol use | Yearly follow up for 10 years
  Participants will be educated on healthy lifestyle habits and alcohol use will be assessed yearly.
Assess hereditary risk through family history review | Yearly follow up for 10 years
  Each participant's family history will be reviewed to make recommendations for screening or genetic testing based on National Comprehensive Cancer Network guidelines.
Assess lifetime breast cancer risk through the Tyrer-Cuzick version 8 breast risk evaluation tool | Yearly follow up for 10 years
  Participants' breast cancer risk will be assessed using the Tyrer-Cuzick breast cancer risk model. Participants will be referred to appropriate clinics if lifetime risk is greater than 20 percent.
Assess 5- year breast cancer risk through the GAIL breast risk evaluation tool | Yearly follow up for 10 years
  Participants' breast cancer risk will be assessed using the National Cancer Institute's GAIL model. Participants will be referred to appropriate clinics if GAIL 5 year risk is greater than 1.7 percent.
Early detection of malignancies through screening | Yearly follow up for 10 years
  Participants will be educated on screening recommendations by the American Cancer Society. Malignancies will be recorded yearly if found by recommended screenings.
Assess changes in fat mass by SOZO measurements | Yearly follow up for 10 years
  Body composition will be assessed yearly by measurements taken from the SOZO device which uses bioimpedance spectroscopy to measure fat mass.
Assess changes in muscle mass by SOZO measurements | Yearly follow up for 10 years
  Body composition will be assessed yearly by measurements taken from the SOZO device which uses bioimpedance spectroscopy to measure muscle mass.

SECONDARY OUTCOMES:
Assess changes in quality of life by the 5-level EuroQol-5D version (EQ-5D-5L) questionnaire | Yearly follow up for 10 years
  Quality of life will be assessed yearly by the EQ-5D-5L questionnaire. Participants' will self-report their health on a scale numbered 0-100. 100 means the best health you can imagine and 0 means the worst health you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Stephenson, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health-Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets will be available upon requests following institutional approval.
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- See also: Education resources — http://www.aicr.org
- See also: Screening guidelines — http://www.cancer.org